CLINICAL TRIAL: NCT05922319
Title: Effects of Training Dose on Computerized Cognitive Training in People With Cognitive Impairment: A Large-population Retrospective Study
Brief Title: Effects of Training Dose on Computerized Cognitive Training in Patients With Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2023027
Record Dates: First submitted 2023-04-02; First posted 2023-06-28 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Impairment, Mild; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cognitive impairment taking computerized cognitive training: The exposures and outcomes were measured repeatedly during the training process for each patient. The outcomes were compared to assess the effect of different exposures (computerized cognitive training with different doses). A mixed effects model was built to solve the random effects of patients.
  Interventions: Other: Computerized cognitive training with different training doses

INTERVENTIONS:
Other: Computerized cognitive training with different training doses — The training dose was defined as training frequency (number of training days per week) and average training duration per training day. The daily dose was divided into 13 categories with an interval of 5 minutes and the training frequency has 7 categories according to the number of training days per week.

SUMMARY:
The goal of this observational study is to explore the optimal dose of computerized cognitive training in patients with cognitive impairment. The main questions it aims to answer are:

* Is there an optimal dose of computerized cognitive training for patients with cognitive impairment?
* Is the optimal dose different in patients in different age populations? Participants enrolled in the study took a reported computerized cognitive training program and the training data were analyzed for exploring the optimal dose.

The researchers will compare the different dose groups to see if there is an optimal dose for the highest improvement in cognitive abilities.

The researchers will additionally compare two age groups (aged younger than 60y or aged 60y and older) to see if the optimal doses in the two groups are different.

DETAILED DESCRIPTION:
Background: Computerized Cognitive Training (CCT) is a form of digital therapeutics that uses computerized cognitive tasks to train patients with cognitive impairment caused by various neurological or psychiatric diseases. CCT has been shown to slow the progression of cognitive impairment in early-stage dementia, particularly in working memory. However, there is a lack of research on the optimal training dose for people with cognitive impairment. Previous meta-analyses have explored the types, delivery methods, and training dose of cognitive training in healthy older adults and those with dementia risk factors, but not in those with cognitive impairment.

Objectives: The study aimed to explore the dose-response relationship of CCT and estimate the optimal daily and weekly dose for people with cognitive impairment.

Participants and methods: the study is a retrospective cohort study and will enroll 21845 patients with cognitive impairment. The exposures in the study are different doses of cognitive training in a week and the outcome is the improvement in cognitive abilities in a week. The weeks with the same training dose of different patients will be classified into one group of exposure. The mixed effects model will be used to estimate the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cognitive impairment.
* Patients who took computerized cognitive training in 2017-2022.
* age ≥ 40 years
* Training duration ≥ 2 weeks

Exclusion Criteria:

* with moderate to severe dementia, cancer, unstable systemic diseases, or psychiatric diseases

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are outpatients who took a reported computerized cognitive training program at home in 2017-2022 in China.
Sampling Method: Non-Probability Sample
Enrollment: 21845 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive abilities between the adjacent weeks | At the end of each week through the study completion (up to 5 years)
  Cognitive ability is measured on the final day of training each week. The cognitive ability throughout a week is calculated based on the overall performance of cognitive training. The overall training performance is an averaged performance integrating the performance of all cognitive training tasks targeting different cognitive domains (e.g., thinking, memory, perception, attention, executive function). The performance of a certain training task is standardized according to normative scores from 0 to 100. Change in cognitive abilities is quantified as the disparity of cognitive abilities between the adjacent weeks (the measurement will be executed everyweek repeatedly).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, M.D., Ph.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China